CLINICAL TRIAL: NCT02779049
Title: The Pathogenic Role and Diagnostic Implication of Program Cell Death Receptor 1 Expressed on T Cells in Mycobacterium Avium Complex Lung Disease
Brief Title: Program Cell Death Receptor 1 in Mycobacterium Avium Complex Lung Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201407079RIND
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Mycobacterium Avium
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- MAC-LD: patients with MAC-LD Do Blood examination
  Interventions: Other: Blood examination
- Control: controls without NTM or tuberculosis infection Do Blood examination
  Interventions: Other: Blood examination
- Tuberculosis infection: patients with tuberculosis infection which diagnosis by culture or typical pathology Do Blood examination
  Interventions: Other: Blood examination
- MAC colonization: patients with MAC pulmonary colonization by American Thoracic Society guideline Do Blood examination
  Interventions: Other: Blood examination

INTERVENTIONS:
Other: Blood examination — blood sampling

SUMMARY:
1. To understand the components of PBMC in MAC-LD patients, including T cells, B cells, nature killer cells, and monocyte.
2. To confirm the phenomenon of reduced PBMC response in MAC-LD patients
3. To study the proportion of apoptosis and PD-1 expression in T cells among MAC-LD patients, MAC colonizers, patients with tuberculosis, and healthy controls.
4. To study the apoptosis and PD-1/PD-L1 expression in T cells/macrophage from bronchial lavage among MAC-LD patients, MAC colonizers, patients with tuberculosis,
5. To examine the PD-1 gene polymorphism and the correlation with MAC-LD.

DETAILED DESCRIPTION:
Background: Nontuberculous mycobacteria Lung disease (NTM-LD) becomes an important clinical concern, because its incidence has increased over the last decade. Mycobacterium avium complex (MAC) is the most common responsible species for NTM-LD in Taiwan. The clinical relevance of MAC in sputum is, however, only 35~42% because it exists in the environment ubiquitously. According to the guideline of the American Thoracic Society, the diagnosis of MAC-LD is based on clinical, radiographic, and mycobacteriology criteria which require two or more positive sputum cultures for MAC. The major limitation of mycobacterial culture is the long turn-around-time, usually 2-4 weeks. In addition, both mycobacterial culture and nucleic acid amplification test cannot discriminate true MAC infection and colonization because airway colonization of MAC is not uncommon. Therefore, diagnosis of MAC-LD remains a big challenge in clinical practice, and rapid and accurate diagnostic test should be developed.

Beyond the contemporary diagnostic criteria, the host immune response in NTM disease has recently been proposed to help diagnosis. Inflammatory markers may represent host response and discriminate MAC infection from colonization. But inflammatory markers can be influenced by infection other than MAC infection. By contrast, lymphocyte response to antigen stimulation may be more specific in diagnosis. In our preliminary results, in-vitro response of peripheral blood mononuclear cell (PBMC) is lower in MAC-LD than healthy controls. The underlying mechanism responsible for the reduced PBMC response in MAC-LD is not fully understood. In previous studies conducted in tuberculosis patients, interaction between programmed cell death ligand-1 (PD-L1) from dendritic cells and programmed cell death-1 (PD-1) in T cells leads to apoptosis or anergy of T lymphocyte and thus suppresses cellular immunity. Therefore, it is possible that similar alteration in immune response also occurs in patients with MAC-LD and correlates with the PBMC response as well as disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* MAC lung disease: Diagnosis is based on the guidelines by American Thoracic Society. In brief, there should be pulmonary symptoms, comparable findings in chest image and appropriate exclusion other possible causes as well as meeting the microbiology criteria.
* MAC pulmonary colonizers: Those without fulfilling the diagnostic criteria but having at least one set of positive sputum for MAC are defined.
* Healthy controls:
* Active tuberculosis group: patients with pulmonary tuberculosis diagnosed by positive respiratory culture

Exclusion Criteria:

* Patients who have acquired immunodeficiency syndrome

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Mycobacterium avium complex lung disease
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percent of disease progression | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided